CLINICAL TRIAL: NCT04333030
Title: INFO-AIDE-TABAC Study on the Level of Information on the Risks Related to Tobacco of Persons Consulting in Psychiatry and on Access to Aids in Case of Smoking, Comparing With Persons Consulting in Diabetology or in Addictology
Brief Title: Study on the Level of Information on the Risks Related to Tobacco of Persons Consulting in Psychiatry and on Access to Aids in Case of Smoking, Comparing With Persons Consulting in Diabetology or in Addictology
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Nadia YOUNES, principal investigator, Versailles Hospital
Other Study IDs: P19/12_info_aide_tabac
Record Dates: First submitted 2020-02-28; First posted 2020-04-03 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Consumption, Tobacco
MeSH Terms: conditions — Tobacco Use | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psychiatry: patients who come for psychiatric consultation
  Interventions: Other: questionnaire
- addictology (other than tabacco): patients who come for addictology consultation
  Interventions: Other: questionnaire
- endocrinology: patients who come for endocrinology consultation
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Tobacco Use and Risk Questionnaire

SUMMARY:
this is an observational study that involves providing a questionnaire to patients consulting in psychiatry, addictology (other than tobacco) and endocrinology to assess their knowledge of tobacco risks and access to smoking cessation aids

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Men and women
* who comes for consultation during the study
* Psychiatry on CMP or HDJ, regardless of diagnosis or smoking status
* Endocrinology in consultation or HDJ
* In addictology at CSAPA

Exclusion Criteria:

* Patient unable to complete questionnaire (not speaking French, confused, alcoholics, etc.)
* Refusal to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who come at :
  * Department of Psychiatry for Adults of the Hospital of Versailles of Dr N Bazin (André Mignot in Chesnay): CMP (Centre Médico-psychologique), HDJ (Day Hospital).
  * Endocrinology service of Dr JP Beressi of the Hospital of Versailles (André Mignot in Chesnay): consultation, HDJ
  * Addictology service CSAPA (Espace Murger) by Dr F Vorspan of the Fernand-Widal Hospital in Paris
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
to Assess the level of information on tobacco-related risks of patients with questionnaire | at the end of study, average 2 month
  to Assess the level of information on tobacco-related risks of patients monitored for psychiatric disorders by comparing them to patients monitored for an addiction other than tobacco or to patients monitored for a chronic disease
to Assess access to smoking cessation aids for smokers and ex-smokers with questionnaire | at the end of study, average 2 month
  to Assess access to smoking cessation aids for smokers and ex-smokers among psychiatric patients compared to smokers and ex-smokers among patients who have been monitored for an addiction other than tobacco or among patients who have been monitored for a chronic disease (endocrine).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Ferdinand Widal, Paris